CLINICAL TRIAL: NCT07399704
Title: Open-label Study to Evaluate the Long-term Safety, Tolerability, Pharmacokinetics and Efficacy of Nizubaglustat (AZ-3102) in Patients With GM2 Gangliosidosis or Niemann-Pick Type C Disease, With or Without Previous Administration of Miglustat
Brief Title: A Study to Evaluate the Safety and Efficacy of Nizubaglustat (AZ-3102) in Patients With GM2 Gangliosidosis or Niemann-Pick Type C Disease
Acronym: PRISMA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azafaros A.G. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA-001-5A2-02
Record Dates: First submitted 2025-12-17; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: GM2 Gangliosidosis; Niemann-Pick Type C Disease
Keywords: Nizubaglustat
MeSH Terms: conditions — Gangliosidoses, GM2; Niemann-Pick Disease, Type C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental): Arms (both cohorts 1 and 2): Nizubaglustat (AZ-3102)
  Interventions: Drug: AZ-3102

INTERVENTIONS:
Drug: AZ-3102 — Daily oral intake of AZ-3102 dispersible tablets

SUMMARY:
This open-label study aims to gather long-term safety, tolerability, PK, biomarker, and clinical efficacy data relating to daily administration of Nizubaglustat in participants previously enrolled in the Phase 2 RAINBOW study (Cohort 1). In addition, the study aims to assess safety, clinical, and biochemical impact of transitioning NPC disease patients to Nizubaglustat after prior treatment with stable, full-dose Miglustat (Cohort 2).

DETAILED DESCRIPTION:
This is a multicenter, open-label study to assess the safety, tolerability, PK, PD, and efficacy of Nizubaglustat in male or female patients with late-infantile or juvenile onset GM2 gangliosidosis or NPC disease in two cohorts:

* Cohort 1: Patients who previously took part in Phase 2 Study AZA-001-5A2-01 (RAINBOW) and wish to continue in this open-label study
* Cohort 2: Approximately 10 patients with NPC disease, aged ≥12 years who received full-dose Miglustat for more than 12 months, have stable or worsening disease over the 2 previous clinic visits, and who wish to stop Miglustat treatment and transition to Nizubaglustat.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 (NPC and GM2 patients):

  * Have been randomized into Phase 2 Study AZA-001-5A2-01.

OR

Cohort 2 (NPC patients):

* Be male or female aged ≥12 years
* Have a genetically-confirmed diagnosis of NPC disease
* Have received full-dose Miglustat treatment for at least 12 months and experienced disease stabilization or worsening with treatment over the 2 previous clinic visits. Patients experiencing clinical improvement with Miglustat over the preceding 3 months should not be considered for this study.
* Wish to change treatment to Nizubaglustat for their NPC disease.
* Participants from Phase 2 Study AZA-001-5A2-01 (RAINBOW) who transitioned to Miglustat may be eligible for Cohort 2 if they meet all other criteria.

Participation is supported and deemed beneficial by the Principal Investigator. Be willing and able to be evaluated for all protocol assessments. The participant, parent, and/or legal guardian can read, understand, and sign the informed consent form. Where appropriate, assent will also be sought for participants who have not reached the age of majority.

Exclusion Criteria:

* A positive serum pregnancy test (only tested for women of childbearing potential).
* Female planning to breastfeed during the study.
* Any medical event/condition that prevents participation in the study based on the judgment of the Principal Investigator.
* Participation in another interventional or non-interventional study or early access program.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2030-04-15 (Estimated); Study Completion 2030-08-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in treatment-emergent adverse events (TEAEs) | Through study completion, an average of 4 years
  Incidence and severity of all Adverse Events related to study drug treatment, study discontinuation or death
Change from baseline in electrocardiogram (ECG) | Through study completion, an average of 4 years
  ECG read out Normal, Abnormal, Not Clinically Significant, Abnormal, Clinically Significant and Not Done.
Change from baseline in seizures | Through study completion, an average of 4 years
  Seizure duration (minutes) as per the seizure diary.
Change from baseline in seizures | Through study completion, an average of 4 years
  Seizure frequency (number) as per seizure diary.
Maximum observed plasma concentration (Cmax) | Baseline , Month 1 (Cohort 2 only) and Month 6
Time to Cmax (Tmax) | Baseline, Month 1 (Cohort 2 only) and Month 6
Concentration at trough (Ctrough) | Baseline, Month 1 (Cohort 2 only) and Month 6
Area under the plasma concentration-time curve from the time of dosing (zero) to 24 hours post-dose | Baseline, Month 1 (Cohort 2 only) and Month 6

SECONDARY OUTCOMES:
Change from Baseline in the concentrations of Glucosylceramide (GlcCer) C16:0; C18:0 | Baseline, Month 1 (Cohort 2 only) and Month 6
Change from Baseline in the concentrations of Neurofilament light chain (NfL) | Through study completion, an average of 4 years
For GM2 gangliosidosis patients: Change from Baseline in the concentrations of Monosialoganglioside GM2 (GM2) | Through study completion, an average of 4 years
For GM2 gangliosidosis patients: Change from Baseline in the concentrations of Lyso-monosialoganglioside GM2 | Through study completion, an average of 4 years
For NPC disease patients: Change from Baseline in the concentrations of N-palmitoyl-O-phosphocholine-serine (PPCS) | Through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Associação Hospitalar de Prot à Infância Dr. Raul Carneiro, Água Verde, Curitiba
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto Nacional de Saúde da Mulher, da Criança e do Adolescente Fernandes Figueira, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No